CLINICAL TRIAL: NCT03433690
Title: The Effect of High Intensity Interval Training in Handling Obesity in Children and Adolescents. A Randomized Controlled Trial.
Brief Title: The Effect of HIIT in Handling Obesity in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regionshospital Nordjylland (Other Government)
Responsible Party: Principal Investigator, Tine Caroc Warner, Principal investigator, M.D., Regionshospital Nordjylland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RHN_TCW_01
Record Dates: First submitted 2018-01-25; First posted 2018-02-14 (Actual); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: High Intensity Interval Training; Child Obesity
Keywords: Child Obesity; Adolescents; High Intensity Interval Training; Moderate training
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: Randomized Controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Intensity Interval Training (Experimental): Twelve weeks of High Intensity Interval Training, twice a week, in combination with multidisciplinary treatment at outpatient obesity clinic.
  Interventions: Behavioral: HIIT
- Moderate training (Active Comparator): Twelve weeks of Moderate Training, twice a week, in combination with multidisciplinary treatment at outpatient obesity clinic.
  Interventions: Behavioral: Moderate training

INTERVENTIONS:
Behavioral: HIIT — High Intensity Interval Training for twelve weeks
  Arms: High Intensity Interval Training
Behavioral: Moderate training — Moderate training for twelve weeks
  Arms: Moderate training

SUMMARY:
In this study the investigators wish to investigate whether a short duration High-intensity Interval Training(HIT) is superior to a moderate activity training modus with regards to improving weight-loss, Blood pressure and sleep quality in severely obese children and adolescents also receiving a multidisciplinary treatment regime.

DETAILED DESCRIPTION:
Prevalence of overweight and obesity among children and adolescents are rapidly rising worldwide. Despite the alarming situation, great confusion of how to tackle obesity persists for two main reasons: the condition is much more complex than initially thought, and many aspects regarding pathophysiology remain unrevealed, leading to an insufficient understanding of the disorder. Childhood obesity is, strongly associated with numerous disorders e.g. hypertension, insuline resistance, sleep apnea, depression and many more.

High intensity Interval Training has proven beneficial in treating obesity and comorbidities in adults. The investigators wish to investigate whether twelve weeks of High-intensity Interval Training(HIT) twice a week is superior to a moderate activity training modus for same period of time with regards to improving weight loss, blood pressure and sleep quality, in severely obese children and adolescents also receiving a multidisciplinary treatment regime. Participants are severely obese children and adolescents referred to the outpatient Clinic for treatment of obesity. Participants are randomizid to either moderate training or HIIT. Antropometric measures, blood pressure and sleep quality as measured by sensewear armbands, are done at baseline, after the twelve weeks of training and again one year after inclusion. Participants are monitored with pulse monitors during training sessions to register if training goals are obtained.

ELIGIBILITY:
Inclusion Criteria:

* Iso-BMI > 30 according to the IOTF iso-BMI cut-off points
* Age 8-18 years of age

Exclusion Criteria:

* Weight below iso-BMI 30, according to the IOTF iso-BMI cut-off points
* Mental illness in the child or the parents that complicates attendance at activities.
* Physical limitations or illness that prevent the child from performing exercise
* If participant is not able to perform all 12 weeks of exercise for other reasons.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2015-07-28 (Actual); Primary Completion 2018-01-25 (Actual); Study Completion 2018-01-25 (Actual)

PRIMARY OUTCOMES:
Weight reduction | Twelve months
  In Kg

SECONDARY OUTCOMES:
Blood pressure | At baseline, after twelve weeks training and after twelve months
  24-hour blood pressure Measurements done by spacelaps 90217A
Sleep Quality | At baseline, after twelve weeks training and after twelve months
  Measured by sensewear armbands which is worn for a week at a time

IPD SHARING:
Plan to Share IPD: No